CLINICAL TRIAL: NCT02309476
Title: Manchester Pascal Endpoint Management Laser Treatment of Diffuse Diabetic Macular Oedema (DMO): A Safety and Efficacy Study
Brief Title: Sub-threshold Photocoagulation of Diabetic Macular Oedema
Acronym: MEM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI decided to close the study early as patients with diffused macular oedema without any previous treatment are uncommon.
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Topcon Corporation (Industry); Optos, PLC (Industry)
Responsible Party: Principal Investigator, Emma Columbine, Professor Paulo Stanga, Manchester University NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03018
Record Dates: First submitted 2014-09-29; First posted 2014-12-05 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Macular Oedema
Keywords: diffuse diabetic macular oedema; Pascal; Laser; DMO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- PASCAL Laser, Green Laser 0.75 (Experimental): Barely Visible Pascal laser grid using 532nm "green" wavelength, 0.75 burn-widths-apart. Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: barely visible burn Average power: 100 to 1000 mW Spot spacing: 0.75 burn-widths-apart Distribution: Grid
  Interventions: Device: PASCAL Laser, Green Laser 0.75
- PASCAL Laser, Green Laser 1 burn (Experimental): Barely Visible Pascal laser grid using 532nm "green" wavelength, 1 burn-widths-apart Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: barely visible burn Average power: 100 to 1000 mW Spot spacing: 1 burn-widths-apart Distribution: Grid
  Interventions: Device: PASCAL Laser, Green Laser 1
- PASCAL Laser, 70% Yellow Laser 0.75 (Experimental): Pascal EM at 70% 577nm "yellow" laser grid, 0.75 burn-widths-apart Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: A barely visible burn will be aimed at for the "Landmark" burn and EndPoint Management will be set at 70% to achieve non-visible burns Average power: 100 to 1000 mW Spot spacing: 0.75 burn-widths-apart Distribution: Grid
  Interventions: Device: PASCAL Laser, 70% Yellow Laser 0.75
- PASCAL Laser, 70% Yellow Laser 1 (Experimental): Pascal EM at 70% 577nm "yellow", 1 burn-widths-apart Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: A barely visible burn will be aimed at for the "Landmark" burn and EndPoint Management will be set at 70% to achieve non-visible burns Average power: 100 to 1000 mW Spot spacing: 1 burn-widths-apart Distribution: Grid
  Interventions: Device: PASCAL Laser, 70% Yellow Laser 1
- PASCAL Laser, 40% Yellow Laser 0.75 (Experimental): Pascal EM at 40% 577nm "yellow", 0.75 burn-widths-apart Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: A barely visible burn will be aimed at for the "Landmark" burn and EndPoint Management will be set at 40% to achieve non-visible burns Average power: 100 to 1000 mW Spot spacing: 0.75 burn-widths-apart Distribution: Grid
  Interventions: Device: PASCAL Laser, 40% Yellow Laser 0.75
- PASCAL Laser, 40% Yellow Laser 1 (Experimental): Pascal EM at 40% 577nm "yellow" laser grid, 1 burn-widths-apart Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: A barely visible burn will be aimed at for the "Landmark" burn and EndPoint Management will be set at 40% to achieve non-visible burns Average power: 100 to 1000 mW Spot spacing: 1 burn-widths-apart Distribution: Grid
  Interventions: Device: PASCAL Laser, 40% Yellow Laser 1

INTERVENTIONS:
Device: PASCAL Laser, Green Laser 0.75 — Barely Visible Pascal laser grid using 532nm "green" wavelength, 0.75 burn-widths-apart. Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: barely visible burn Average power: 100 to 1000 mW Spot spacing: 0.75 burn-widths-apart Distribution: Grid
  Arms: PASCAL Laser, Green Laser 0.75
Device: PASCAL Laser, Green Laser 1 — Barely Visible Pascal laser grid using 532nm "green" wavelength, 1 burn-widths-apart. Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: barely visible burn Average power: 100 to 1000 mW Spot spacing: 0.75 burn-widths-apart Distribution: Grid
  Arms: PASCAL Laser, Green Laser 1 burn
Device: PASCAL Laser, 70% Yellow Laser 0.75 — Pascal EM at 70% 577nm "yellow" laser grid, 0.75 burn-widths-apart Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: A barely visible burn will be aimed at for the "Landmark" burn and EndPoint Management will be set at 70% to achieve non-visible burns Average power: 100 to 1000 mW Spot spacing: 0.75 burn-widths-apart Distribution: Grid
  Arms: PASCAL Laser, 70% Yellow Laser 0.75
Device: PASCAL Laser, 70% Yellow Laser 1 — Pascal EM at 70% 577nm "yellow" laser grid, 0.75 burn-widths-apart Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: A barely visible burn will be aimed at for the "Landmark" burn and EndPoint Management will be set at 70% to achieve non-visible burns Average power: 100 to 1000 mW Spot spacing: 1 burn-widths-apart Distribution: Grid
  Arms: PASCAL Laser, 70% Yellow Laser 1
Device: PASCAL Laser, 40% Yellow Laser 0.75 — Pascal EM at 40% 577nm "yellow" laser grid, 0.75 burn-widths-apart Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: A barely visible burn will be aimed at for the "Landmark" burn and EndPoint Management will be set at 740% to achieve non-visible burns Average power: 100 to 1000 mW Spot spacing: 0.75 burn-widths-apart Distribution: Grid
  Arms: PASCAL Laser, 40% Yellow Laser 0.75
Device: PASCAL Laser, 40% Yellow Laser 1 — Pascal EM at 40% 577nm "yellow" laser grid, 0.75 burn-widths-apart Intervention: macular laser grid Number of burns: Full grid 112 burns Spot size: 100micron Duration: 10 ms Exposure: A barely visible burn will be aimed at for the "Landmark" burn and EndPoint Management will be set at 740% to achieve non-visible burns Average power: 100 to 1000 mW Spot spacing: 0.75 burn-widths-apart Distribution: Grid
  Arms: PASCAL Laser, 40% Yellow Laser 1

SUMMARY:
Topcon's Endpoint Management (EM) is a new software from the Pascal® laser which allows us to decrease the intensity of the burns (invisible burns) showing some landmarks with normal intensity so the investigators can see the area which has been treated. The Pascal® system with EM utilizes 577nm laser wavelength compared to the 532nm laser wavelength which was utilized in previous Pascal® laser studies.

This study aims to demonstrate that 577nm Pascal® with EM has the same efficacy and effectiveness as 532nm Pascal® in the treatment of diabetic macular oedema.

DETAILED DESCRIPTION:
Diabetic macular oedema (DMO) remains the most common cause of visual loss in diabetic patients and affects around 29% of diabetic patients with 20 or more years of disease. The Early Treatment Diabetic Retinopathy Study (ETDRS) demonstrated a significant benefit of laser photocoagulation for the treatment of clinically significant macular oedema, reducing the incidence of vision loss by approximately 50% at 3 years' follow-up.

The original ETDRS photocoagulation technique was adopted throughout the world and gradually modified through the years. Despite the great improvements, loss of central vision, paracentral scotoma and decreased color vision are some adverse events that can still occur, mostly caused by the progressive enlargement of the laser scars consequent to the visible burn of conventional laser photocoagulation.

New strategies have been developed for laser treatments that minimize the chorioretinal damage while maintaining at least similar treatment efficacy.

And numerous clinical studies have been conducted with subvisible laser treatments. However, the lack of a visible endpoint makes it difficult for the treating physician to know which retinal areas have been treated in order to avoid retreatment and also to be confident that the desired target tissue had been treated.

Topcon's Endpoint Management (EM) is a new software from the Pascal® laser which allows us to decrease the intensity of the burns (invisible burns) showing some landmarks with normal intensity so the investigators can see the area which has been treated.

The Pascal® system with EM utilizes 577nm laser wavelength compared to the 532nm laser wavelength which was utilized in previous Pascal® laser studies.

This study aims to demonstrate that 577nm Pascal® with EM has the same efficacy and effectiveness as 532nm Pascal®.

ELIGIBILITY:
Inclusion Criteria:

Patient-eligibility

Inclusion criteria:

1. Older than 18 years of age
2. Male or female patients with diabetes mellitus type I or type 2 who meet the WHO or ADA criteria for diabetes
3. Able to give informed consent

Study Eye eligibility

Inclusion criteria:

1. ETDRS visual acuity equivalent to 35 letters or better (Snellen equivalent 20/200 or better)
2. The patient must have non-proliferative diabetic retinopathy (NPDR) with diffuse macular oedema
3. Mean average central retinal thickness at least 300 microns as measured by Deep Range Imaging Optical Coherence Tomography (DRI -OCT) scans
4. Adequate pupil dilatation and clear media to perform wide-field colour, red-free imaging and fundus fluorescein angiography (WF-FFA), wide-field fundus autofluorescence imaging (WF-AF) and DRI-OCT
5. Ability to perform accurate Humphmrey visual field test

Exclusion Criteria:

Patient-eligibility

Exclusion criteria:

1. History of chronic renal failure or renal transplant for diabetic nephropathy
2. Recent (last 6 months) or on-going poor glycaemic control. H1Ac greater than 10.0mg/dL
3. Creatinine greater than 1.2 mg/dL
4. HDL equal to or greater than 40 mg/dL
5. Uncontrolled hypertension. Blood pressure greater or equal to 180/110 mmHg
6. Patient is unavailable for follow-up visits
7. Pregnant women or breast-feeding females

Study Eye eligibility

Exclusion criteria:

1. Lens opacity that could influence vision and results
2. Proliferative Diabetic Retinopathy.
3. Any surgical or non-retinal laser treatment to the study eye within 2 months
4. Narrow drainage angles with raised intraocular pressure and angle closure glaucoma.
5. Planned YAG peripheral iridotomy
6. Previous retinal laser photocoagulation, intraocular drug therapy, or macular laser treatment to treatment eye in last year
7. Vitreomacular traction determined clinically and / or OCT, which in the opinion of the investigator, contributes to macular edema (associated or cause a detachment of the fovea) and prevents the improvement with treatment.
8. Atrophy / scar / fibrosis involving the center of the macula, including evidence of atrophy treated with laser within 200 microns of the FAZ.
9. Any previous ocular condition that may be associated with a risk of macular edema
10. Important known allergies to sodium fluorescein dye used in angiography.

12. Active lid or adnexal infection 13. Planned intra-ocular surgery within one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
reduction of diabetic macular edema (central retinal thickness) within the 6 arms of the study | 12 months
  To compare Green Pascal® laser and Yellow Pascal® laser using EM among 6 groups of participants using Pascal® laser with an application of full grid 112 burns in a single session

SECONDARY OUTCOMES:
Improvement in visual acuity (> 10 letters or two lines in the ETDRS chart) | 12 months
increase in retinal sensitivity within the 6 arms of the study | 12 months
  increase in retinal sensitivity will be assessed with fundus-related perimetry (microperimetry)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Stanga, Principal Investigator — Manchester Royal Eye Hospital
Locations (1):
- Central Manchester Foundation Trust, Manchester, England, United Kingdom